CLINICAL TRIAL: NCT04672889
Title: Use Babyguard® Breast Milk Probiotics to Verify the Authenticity of the Gut-Breast Axis Hypothesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201703031RINC
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Intestinal Bacteria Flora Disturbance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): consume 1 sachet per day for 1 months
  Interventions: Dietary Supplement: Placebo
- Babyguard® Breast Milk Probiotics (Experimental): consume 1 sachet per day for 1 months
  Interventions: Dietary Supplement: Babyguard® Breast Milk Probiotics

INTERVENTIONS:
Dietary Supplement: Placebo — consume 1 sachet per day for 1 months
  Arms: Placebo
Dietary Supplement: Babyguard® Breast Milk Probiotics — consume 1 sachet per day for 1 months
  Arms: Babyguard® Breast Milk Probiotics

SUMMARY:
In order to understand the life history of the breast milk flora, explore its composition, source of strains, and ability to colonize the baby's intestinal environment, to find out strains with the potential of probiotics in breast milk

DETAILED DESCRIPTION:
This is a double-blind and randomized study. After being discharged from the hospital, the subject was notified to consume the Babyguard breast milk probiotic daily for 1 month, and observe whether the mother's stool, breast milk and baby stool samples can find the same strain. The clinical diagnosis items of the bacterial strains of mother feces, breast milk and baby feces samples are evaluated by the doctor.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old, pregnant women with non-high-risk pregnancy risk assessed by obstetricians and gynecologists, healthy mothers and infants with no abnormal obstetric examination results

Exclusion Criteria:

* Pregnant women who have used oral or injectable antibiotics within three months before delivery, or women who need a cesarean section for any reason during pregnancy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Those who are 20 years old and pregnant
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Microflora of mother's feces | 4-6 weeks after the baby is born
  Collect mother's feces for bacterial analysis.The mother's feces use Qiagen stool mini kit to extract DNA, and then use the intestinal bacteria primers to detect the presence of intestinal bacteria in the feces.
Group. B Streptococcus (GBS) screening | 35-37 weeks of pregnancy
  Use sterile cotton sticks for vaginal samples, and then perform Group. B Streptococcus (GBS) screening
The microflora of maternal blood | 4-6 weeks after the baby is born
  Use venous blood to collect 20 ml of mother's blood for bacterial analysis.The mother's blood uses Qiagen DNA isolation mini kit to extract DNA, and then uses intestinal bacteria primers to detect the presence of intestinal bacteria in the blood
Metabolic analysis of maternal urine | 4-6 weeks after the baby is born
  Collect 10 ml of mother's urine for intestinal dysbiosis analysis. Use Qiagen DNA isolation mini kit to extract DNA from the mother's urine, and then use the intestinal bacteria primer to detect the presence of intestinal bacteria in the urine.
Bacteria analysis of breast milk | 4-6 weeks after the baby is born
  Collect 10 ml of breast milk for bacterial phase analysis.Use Qiagen DNA isolation mini kit to extract DNA from breast milk, and then use intestinal bacteria primers to detect whether the breast milk contains intestinal bacteria.
Bacteria analysis of infant feces | 4-6 weeks after the baby is born
  Collect baby feces for bacterial phase analysis.Use Baby feces use Qiagen stool mini kit to extract DNA, and then use intestinal bacteria primers to detect the presence of intestinal bacteria in the feces.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shiang Wu, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan